CLINICAL TRIAL: NCT06080269
Title: To Compare the Effect of Receiving the Technology-based Training Along With the Conventional Therapy to the Conventional Therapy Alone on Executive Functions Among People With Traumatic Brain Injury With Mild to Moderate Cognitive Deficit: A Pilot Randomized Control Trial
Brief Title: To Compare the Effect of Receiving the Technology-based Training Along With the Conventional Therapy to the Conventional Therapy Alone on Executive Functions Among People With Traumatic Brain Injury With Mild to Moderate Cognitive Deficit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-21-857
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury Rehabilitation; Technology based intervention; Cognitive retraining; Executive functions
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Masking Description: No blinding was done hence its a open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The participants in the intervention arm will be receiving technology based training along with the conventional therapy
  Interventions: Device: technology based intervention along with conventional therapy
- Control arm (Active Comparator): The participants in the control arm will be receiving the regular conventional therapy program
  Interventions: Other: conventional therapy alone

INTERVENTIONS:
Device: technology based intervention along with conventional therapy — Technology based intervention are training session given to the participants through devices which has software installed to train cognitive functions for patients with cognitive deficit.
  Arms: Intervention arm
Other: conventional therapy alone — Participants in the control group will receive only conventional therapy
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to compare the effect of receiving the technology-based training along with the conventional therapy to the conventional therapy alone on executive functions among people with traumatic brain injury with mild to moderate cognitive deficit.

It aims to answer:

* If there is significant improvement in executive function skills among people with traumatic brain injury receiving technology-based training along with conventional therapy when compared to people with traumatic brain injury receiving conventional therapy alone.
* To see if the demographic variable has any effect on the cognitive improvement

Participants will in the intervention group will be given 45 minutes of extra training session using technology along with their usual rehabilitation session.

And Participants in the control group will be receiving the usual rehabilitation sessions.

Researchers will compare the changes in the outcome measures between the intervention and control group to see if the technology-based training along with conventional therapy had significant effect on executive skills among people with traumatic brain injury.

DETAILED DESCRIPTION:
Cognitive deficit following traumatic brain injury is one of the important consequences affecting the individual's quality of life. Various cognitive intervention strategies are in practice and the use of technology-based cognitive interventions are into current practice. This study is a Pilot Randomized Control Trial which aims to compare the effect of receiving the technology-based training along with the conventional therapy to the conventional therapy alone on executive functions among people with traumatic brain injury with mild to moderate cognitive deficit. This study will be done in Qatar Rehabilitation Institute, Hamad Medical Corporation, Doha, Qatar. People with traumatic brain injury with mild to moderate cognitive deficit (MMSE>10 and <23), between the age group of 18 to 60 years, no previous history of head trauma and willing to comply with cognitive rehabilitation program will be recruited for this study. The investigators will be explaining the details of the study to the participants and the participants who are willing to take part in the study had to give their consent by signing the consent sheet. After which they will be randomized in either intervention or control group through envelop concealment method. After randomization, the participants will be assessed using the outcome measures such as MMSE, Cognitive FIM and Executive function performance test (EFPT), one day before the start of the intervention. Participants in the intervention group will be receiving extra 45 min of technology based cognitive circuit training using MYRO, BITS and Cognitive Rehametrics in addition to the conventional therapy and participants in the control group will be receiving the regular conventional therapy alone. As a part of conventional therapy, participants will be receiving an hour of occupational therapy which focuses on all aspects of the deficit. For cognitive deficit, the participants will be receiving traditional method of training that includes paper pencil task, tabletop activities, performance-based activities and computer-based activities. Participants in both the groups will be receiving the sessions 5 times a week for 6 weeks. At the end of 6 weeks, all the participants in both groups will be assessed using the outcome measures, and the data will be collated, coded and entered in an excel sheet. The coded data will be sent for the statistical analysis.

Baseline characteristics will be presented as means±SD or median for continuous data, and as frequencies and associated percentages for categorical parameters. The statistical P value for change from baseline for quantitative outcomes will be calculated with a paired test or Wilcoxon signed rank test, and the P value for the difference between intervention and control groups will be calculated using unpaired t or Mann Whitney U tests appropriate.

Associations between two or more qualitative variables will be assessed using Chi-square (χ2) or Fisher Exact tests as appropriate. Relationship between two quantitative variables (age, EFPT, FIM scores etc.) will be examined using Pearson's or Spearman's correlation coefficients. All primary efficacy analyses will be performed on the intent-to-treat (ITT) population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with traumatic brain injury i.e damage to the brain resulting from external mechanical force, such as rapid acceleration or deceleration, impact, blast waves, or penetration by a projectile
2. Adults aged between 18 and 60 years old
3. No previous history of head trauma
4. With MMSE score >10 and < 23 (people with mild to moderate cognitive deficit)
5. Ability to give consent and willingness to comply with cognitive rehabilitation program.

Exclusion Criteria:

1. Pre-existing chronic illness that causes neurological symptoms or complications such as congenital disorder, history of stroke, tumor, brain infection or any other previous disorder due to brain damage affecting the cognition.
2. History of any psychiatry disorders which affects the cognitive functions such as schizophrenia, bipolar disorder etc.
3. Those who cannot follow basic simple instruction or comprehend simple commands

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Executive Function Performance Test (EFPT) | 2 times, one before the intervention and one after 6 weeks
  It's a performance-based assessment that measures the executive functions. It has score ranging from 0 to 50, where higher the score higher is the executive skills

SECONDARY OUTCOMES:
Cognitive functional independence measure scale (CogFIM) | 2 times, one before the intervention and one after 6 weeks
  Functional Independence measure is a test that evaluated the participants independence in functional activities and CogFIM measure the independence in social cognition. The score ranges from 0 to 35, where higher the scores indicates higher is the social cognitive skills.
Mini Mental State Examination -2 (MMSE-2) | 2 times, one before the intervention and one after 6 weeks
  It's a tool to measure the general cognitive functions of the participants. This tool can be used as a screening tool and as an outcome tool. The score ranges from 0 to 30 where higher the score higher is the general cognition.

CONTACTS AND LOCATIONS:
Locations (1):
- Qatar Rehabilitation Institute, Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Patients' identity will not be revealed. The data will be coded and will be sent to other researchers for analysis purpose.